CLINICAL TRIAL: NCT01726257
Title: Prospective, Multicenter, Single Arm Safety and Effectiveness Study of Endovascular Abdominal Aortic Aneurysm Repair Using the Nellix® System: A Pivotal and Continued Access Study
Brief Title: Safety and Effectiveness Study of Endovascular Abdominal Aortic Aneurysm Repair Using the Nellix® System
Acronym: EVAS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0008
Record Dates: First submitted 2012-10-19; First posted 2012-11-14 (Estimated); Results first posted 2024-11-06 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: Infrarenal; Abdominal; Aortic; Aneurysm; AAA; Endologix; EVAS; EndoVascular; Sealing; System
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Nellix System (Experimental): Nellix Endovascular Aneurysm Sealing System is the only arm for this study. This is a single arm study.
  Interventions: Device: Nellix System

INTERVENTIONS:
Device: Nellix System — Subjects in this study will receive a Nellix Endovascular Sealing System as part of their intervention.

SUMMARY:
The objective of this study is to assess the safety and effectiveness of the Endologix Nellix® System for the endovascular repair of infrarenal abdominal aortic aneurysms (AAA).

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of the Nellix System among a wide range of physicians and in consecutively enrolled subjects to assess outcomes generalizability. Following appropriate government and ethics committee/IRB approval the Nellix® EndoVascular Sealing System will be implanted into eligible patients who are adequately informed and have consented to join the study. Enrolled patients will undergo a high resolution, contrast-enhanced computed tomography angiography (CT) scan of the relevant aortic and aortoiliac vasculature within three months of the scheduled procedure and at specified follow-up intervals post-implantation. Follow-up visits will occur at 30 days, 6 months, and annually to 5 years to assess aneurysm morphology, the status of the implanted devices, and relevant laboratory test results.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old;
* Informed consent understood and signed;
* Patient agrees to all follow-up visits;
* Have AAA with sac diameter ≥5.0cm, or ≥4.5 cm which has increased by >1.0cm in the past year.
* Anatomic eligibility for the Nellix System per the instructions for use:
* Adequate iliac/femoral access compatible with the required delivery systems (diameter ≥6 mm);
* Aneurysm blood lumen diameter ≤60mm;
* Most caudal renal artery to aortoiliac bifurcation length ≥100mm;
* Proximal non-aneurysmal aortic neck: length ≥10mm; lumen diameter 18 to 32mm; angle ≤60° to the aneurysm sac;
* Common iliac artery lumen diameter between 9 and 35mm with blood lumen diameter ≤35mm;
* Ability to preserve at least one hypogastric artery.

Exclusion Criteria:

* Life expectancy <2 years;
* Psychiatric or other condition that may interfere with the study;
* Participating in enrollment of another clinical study
* Known allergy to device any device component;
* Coagulopathy or uncontrolled bleeding disorder;
* Ruptured, leaking or mycotic aneurysm;
* Serum creatinine level >2.0mg/dL;
* CVA or MI within three months of enrollment/treatment;
* Aneurysmal disease of the descending thoracic aorta;
* Clinically significant infrarenal mural thrombus (>5mm thickness over >50% circumference);
* Connective tissue diseases (e.g., Marfan Syndrome)
* Unsuitable vascular anatomy;
* Pregnant (females of childbearing potential only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Carpenter, MD, Principal Investigator — Cooper Hospital, Camden, NJ
Locations (30):
- United States (27):
  - Tucson Medical Center, Tucson, Arizona
  - VA San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Christiana Care Hospital, Newark, Delaware
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Baptist Hospital of Miami, Miami, Florida
  - Sacred Heart, Pensacola, Florida
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Bay State Hospital, Springfield, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Minneapolis Hospital, Minneapolis, Minnesota
  - St. Vincent Heart and Vascular Center of Montana, Billings, Montana
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Cooper Hospital, Camden, New Jersey
  - Carolinas Health Care, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Heart and Vascular Institue, Pittsburgh, Pennsylvania
  - St. Luke's Medical Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Scott & White Healthcare System, Temple, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Froedtert Memorial Lutheran Hospital (Medical College of Wisconsin), Milwaukee, Wisconsin
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany
- Rijnstate Hospital, Arnhem, Netherlands
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Kisis K, Krievins D, Naskovica K, Gedins M, Savlovskis J, Ezite N, Lietuvietis E, Zarins K. Quality of life after endovascular abdominal aortic aneurysm repair: nellix sac-anchoring endoprosthesis versus open surgery. Medicina (Kaunas). 2012;48(6):286-91. PMID 22885361
- [Background] Krievins DK, Holden A, Savlovskis J, Calderas C, Donayre CE, Moll FL, Katzen B, Zarins CK. EVAR using the Nellix Sac-anchoring endoprosthesis: treatment of favourable and adverse anatomy. Eur J Vasc Endovasc Surg. 2011 Jul;42(1):38-46. doi: 10.1016/j.ejvs.2011.03.007. Epub 2011 Apr 15. PMID 21497521
- [Derived] Carpenter JP, Lane JS 3rd, Trani J, Hussain S, Healey C, Hashemi H, Cuff R; Nellix Investigators. Proper technical procedures improved outcomes in a retrospective analysis of EVAS FORWARD IDE trial 3-year results. J Vasc Surg. 2020 Sep;72(3):918-930.e2. doi: 10.1016/j.jvs.2019.11.039. Epub 2020 Feb 5. PMID 32035772
- [Derived] Carpenter JP, Lane JS 3rd, Trani J, Hussain S, Healey C, Buckley CJ, Hashemi H, Cuff R; Nellix Investigators. Refinement of anatomic indications for the Nellix System for endovascular aneurysm sealing based on 2-year outcomes from the EVAS FORWARD IDE trial. J Vasc Surg. 2018 Sep;68(3):720-730.e1. doi: 10.1016/j.jvs.2018.01.031. Epub 2018 Mar 31. PMID 29609994
- [Derived] Carpenter JP, Cuff R, Buckley C, Healey C, Hussain S, Reijnen MM, Trani J, Bockler D; Nellix Investigators. Results of the Nellix system investigational device exemption pivotal trial for endovascular aneurysm sealing. J Vasc Surg. 2016 Jan;63(1):23-31.e1. doi: 10.1016/j.jvs.2015.07.096. Epub 2015 Oct 21. PMID 26482997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 180 subjects will be enrolled at a maximum of 30 sites in the EU, and US in the Primary Investigation. This includes up to 30 Roll-in subjects and up to 150 patients in the Intent to Treat Pivotal Cohort. At enrollment closure for the Primary Investigation, an Extended Investigation will commence at these sites to enroll up to 250 additional subjects under continued access provisions. The protocol allowed up to 430 total subjects, however, the actual enrollment total was 333.
Groups:
- Pivotal Cohort (ITT): The Intention to Treat Pivotal Cohort includes up to 150 subjects will be enrolled at a maximum of 30 sites in the US and the EU.This includes the statistically justified sample size of 132 plus an allowance for deviations from assumptions.
- Roll-In Cohort: One (1) roll-in subject may be enrolled per site, therefore a maximum of 30 enrolled in the study, to allow for Investigator(s) to receive additional training on the Nellix System. Any roll-in subjects will be screened, consented, treated and followed identically to the main study cohort.However, the roll-in cohort of this study will be evaluated separately.
- Continued Access Cohort: Up to 250 patients will be enrolled into the Extended Investigation based on an enrollment rate of 0.5 patients per site per month and an estimated 20 months from the close of enrollment in the Primary Investigation. Enrollment in Extended Investigation (continued access) phase will be limited to the 27 US sites only as the Nellix System is commercially available to the three participating European sites.
Period: Overall Study
Arm/Group | Pivotal Cohort (ITT) | Roll-In Cohort | Continued Access Cohort
Started | 150 | 29 | 154
Completed | 86 | 8 | 75
Not Completed | 64 | 21 | 79

BASELINE CHARACTERISTICS:
Groups:
- Pivotal Cohort: Subject Demographics for the Pivotal cohort
- Roll-In Cohort: Subject Demographics for the Roll-in cohort
- Continued Access Cohort: Subject Demographics for the Continued Access cohort
- Total: Total of all reporting groups
Arm/Group | Pivotal Cohort | Roll-In Cohort | Continued Access Cohort | Total
Number analyzed (Participants) | 150 | 29 | 154 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8) | 72 (10) | 73 (7) | 73 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 13 | 21
  Male | 142 | 29 | 141 | 312
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 140 | 25 | 141 | 306
  Race: Non-Caucasian | 10 | 4 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Events at 30 Days
Description: Major Adverse Events = all-cause death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, stroke, and blood loss >1,000cc
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal Cohort | Roll-In Cohort | Continued Access Cohort
Number analyzed (Participants) | 150 | 29 | 154
Participants | 4 | 1 | 2

2. Primary Outcome: Treatment Success at 1 Year
Description: Procedural technical success and the absence of aneurysm rupture, conversion to open surgical repair, Type I endoleak at 12 months, Type III endoleak at 12 months, aneurysm enlargement, secondary procedure for resolution of endoleak (Type I or III), limb occlusion, migration, aneurysm sac expansion and/or a device defect.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal Cohort (ITT) | Roll-In Cohort | Continued Access Cohort
Number analyzed (Participants) | 134 | 26 | 109
Participants | 126 | 22 | 94

ADVERSE EVENTS:
Time Frame: All serious and non-serious events within 30 days, at 6 months, and annually to 5 years
Arm/Group | Pivotal Cohort (ITT) | Roll-In Cohort | Continued Access Cohort
All-Cause Mortality (participants affected / at risk) | 1/150 | 0/29 | 1/154
Serious Adverse Events (participants affected / at risk) | 26/150 | 5/29 | 37/154
Other Adverse Events (participants affected / at risk) | 38/150 | 7/29 | 40/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pivotal Cohort (ITT) (N=150) | Roll-In Cohort (N=29) | Continued Access Cohort (N=154)
Bleeding/Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (4)
Bowel (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiac (Cardiac disorders) | 7 (7) | 0 (0) | 5 (5)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Miscellaneous (General disorders) | 2 (6) | 2 (2) | 4 (4)
Nellix Device (Product Issues) | 0 (0) | 0 (0) | 10 (11)
Neurological (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 4 (7)
Renal (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (1)
Surgical Site Wound (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Urogenital (Renal and urinary disorders) | 4 (4) | 1 (1) | 3 (3)
Vascular (Vascular disorders) | 5 (5) | 2 (2) | 14 (19)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pivotal Cohort (ITT) (N=150) | Roll-In Cohort (N=29) | Continued Access Cohort (N=154)
Bleeding/Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Bowel (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiac (Cardiac disorders) | 8 (8) | 1 (1) | 1 (1)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0)
Miscellaneous (General disorders) | 11 (15) | 3 (3) | 16 (25)
Nellix Device (Product Issues) | 1 (1) | 0 (0) | 1 (1)
Neurological (Nervous system disorders) | 5 (6) | 0 (0) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (6)
Renal (Renal and urinary disorders) | 6 (7) | 0 (0) | 2 (2)
Surgical Site Wound (Surgical and medical procedures) | 13 (15) | 1 (1) | 5 (5)
Urogenital (Renal and urinary disorders) | 4 (5) | 1 (1) | 5 (5)
Vascular (Vascular disorders) | 4 (4) | 0 (0) | 10 (11)
Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT01726257/Prot_SAP_000.pdf